CLINICAL TRIAL: NCT04793412
Title: Cochlear Implantation in Children With Asymmetric Hearing Loss or Single-Sided Deafness Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Louis Children's Hospital (Other); University of Southern California (Other); Children's Hospital of Philadelphia (Other); Hearts for Hearing (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202007142
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Asymmetric Hearing Loss; Single-sided Deafness; Unilateral Deafness
Keywords: hearing loss; cochlear implant
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Intervention Model Description: The study is conducted as a multicenter, prospective, two-phase clinical trial, evaluating the efficacy and safety of cochlear implantation in children with asymmetric hearing loss (AHL) or single-sided deafness (SSD). A hearing aid (HA) phase occurs over a minimum of 4 mos prior to obtaining a cochlear implant (CI). A CI phase occurs over the 15-month period after initial activation of the CI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AHL/SSD (Experimental): Children with asymmetric hearing loss or single-sided deafness
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — Cochlear implantation of a device from one of the three manufacturers available in the US.

SUMMARY:
This is a two-phase study that compares performance growth pre-implant with current hearing aid (HA) technology versus post-implant with a cochlear implant (CI) in children with either asymmetric hearing loss (AHL) or single-sided deafness (SSD). Post-implant performance with a CI alone is expected to outperform pre-implant performance with a HA. The study also evaluates the effectiveness of bimodal hearing defined as a CI in the poor ear and a HA in the better ear for AHL or a CI in the poor ear and normal hearing in the better ear for SSD compared to pre-implant performance. The study examines factors contributing to CI outcomes.

DETAILED DESCRIPTION:
The study is conducted as a multicenter, prospective, two-phase clinical trial, evaluating the efficacy and safety of cochlear implantation in children with asymmetric hearing loss (AHL) or single-sided deafness (SSD). A hearing aid (HA) phase occurs over a minimum of 4 mos prior to obtaining a cochlear implant (CI). A CI phase occurs over the 15-month period after initial activation of the CI. The AHL/SSD groups are tested for change in performance pre- to post-implant. Investigators also collect longitudinal data over 12 months (matching the 3 to 15 month post-implant timeframe) from normal hearing (NH) participants to provide additional information about outcome trajectory due to development alone. The NH participants are matched to AHL/SSD participants on age, gender and parent education. Post-implant performance with a CI alone is expected to outperform pre-implant performance with a HA. The study evaluates the effectiveness of bimodal hearing defined as a CI in the poor ear and a HA in the better ear for AHL or a CI in the poor ear and normal hearing in the better ear for SSD compared to pre-implant performance. The study examines factors contributing to CI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 4 ys of age and up to 14 yrs, 11 mos of age and able to complete all investigational procedures.
* Parents and child fluent in English. Parents desire bilateral hearing for their child, are willing to comply with study requirements, including the pre-implant HA phase, and are able to provide informed consent.
* Poor ear (AHL/SSD): PTA at .5, 1, 2 kHz > 70 dB HL; Aided CNC word recognition score at 60 dB SPL < 40%; SPHL duration ≥ 6 mos and ≤ 10 yrs at time of CI surgery; If > 5 yrs of age, evidence of non-congenital SPHL onset (e.g., passed newborn hearing screening); If ≤ 5 yrs of age, no restrictions on SPHL onset.
* Better ear
* AHL: PTA at .5, 1, 2, 4 kHz > 25 and ≤ 60 dB HL; Aided CNC word score at 60 dB SPL ≥ 55%; Currently using a HA; Stable hearing for the past 6-mo period. "Stable" is defined as thresholds that have not declined by more than 20 dB at three or more octave-interval audiometric frequencies.
* SSD: PTA at .5, 1, 2, 4 kHz ≤ 25 dB HL; CNC word score at 60 dB SPL ≥ 70%; Stable hearing for the past 6-mo period.
* Both ears of NH participants: PTA at .5, 1, 2, 4 kHz ≤ 25 dB HL.
* To continue with cochlear implantation and into the CI phase of the study: Indication, via imaging, of a normal cochlear nerve and of cochlear anatomy in the ear to be implanted that allows full insertion of the electrode array. Imaging modality is at the discretion of the surgeon. In addition, better ear hearing must be stable throughout the HA phase.

Exclusion Criteria for AHL/SSD Participants:

* Medical condition that contraindicates surgery; Actively using an implantable device in the ear to be implanted; Inability to complete study procedures; Unrealistic expectations related to the benefits and limitations of implantation; Unwillingness or inability to comply with all investigational requirements.
* Exclusions for cochlear implantation and the CI phase of the study: Cochlear malformation or obstruction that would preclude full insertion of the electrode array in the ear to be implanted; Abnormal cochlear nerve in the ear to be implanted; Hearing loss of neural or central origin.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Poor ear alone word recognition in quiet from Pre-Implant to 12 months post-implant | Pre-Implant and 12 months post-implant
  Poor ear alone CNC monosyllabic word recognition in quiet with the CI alone compared to pre-implant with a HA.
Change in Bimodal speech understanding in noise from Pre-Implant to 15 months post-implant | Pre-implant and 15 months post-implant
  Speech reception thresholds (SRTs) for understanding words in noise in the bimodal condition (CI + HA for AHL; CI + NH ear for SSD) post-implant compared to the pre-implant best aided condition.
Post-implant bimodal vs better ear alone speech understanding in noise | 15 months post-implant
  Post-implant speech reception thresholds (SRTs) for understanding words in noise in the bimodal condition (CI + HA for AHL; CI + NH ear for SSD) compared to the better ear alone condition.
Change in pre-implant trajectory of Bimodal speech understanding in noise over time to post-implant trajectory over time | 5 visits pre-implant over a minimum of 4 months and the 3, 6, 9, 12, and 15 month post-implant visits
  The trajectory of speech reception thresholds (SRT) for understanding noise throughout the CI Phase (5 visits post-implant) in the bimodal condition is compared to the trajectory throughout the HA Phase (5 visits pre-implant) in the best aided condition.

SECONDARY OUTCOMES:
Change in Poor ear alone audibility from Pre-Implant to 12 months post-implant | Pre-implant and 12 months post-implant
  FM tone sound field threshold levels in the poor ear alone with a CI compared to pre-implant threshold levels with a HA
Change in Bimodal sound localization from Pre-Implant to 15 months post-implant | Pre-implant and 15 months post-implant
  RMS error scores for a sound localization task in the bimodal condition (CI + HA for AHL; CI + NH ear for SSD) post-implant compared to the pre-implant best aided condition.
Change in Bimodal soft speech understanding from Pre-Implant to 12 months post-implant | Pre-implant and 12 months post-implant
  CNC monosyllabic word recognition at a soft level in the bimodal condition (CI + HA for AHL; CI + NH ear for SSD) post-implant compared to the pre-implant best aided condition.
Change in PedsQL-MFS ratings from Pre-Implant to 15 months post-implant | Pre-implant and 15 months post-implant
  Questionnaire completed by parents and participants (when age appropriate). Ratings post-implant are compared to pre-implant ratings.
Change in SSQ ratings from Pre-Implant to 15 months post-implant | Pre-implant and 15 months post-implant
  Questionnaire completed by parents and participants (when age appropriate). Ratings post-implant are compared to pre-implant ratings.
Change in HEAR-QL ratings from Pre-Implant to 15 months post-implant | Pre-implant and 15 months post-implant
  Questionnaire completed by parents and participants (when age appropriate). Ratings post-implant are compared to pre-implant ratings.
Post-implant bimodal vs better ear alone sound localization | 15 months post-implant
  Post-implant RMS error scores for the sound localization task are compared in the bimodal condition to the better ear alone condition.
Post-implant bimodal vs better ear alone soft speech understanding | 12 months post-implant
  Post-implant word recognition scores at soft levels are compared in the bimodal condition to the better ear alone condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jill B Firszt, PhD, Principal Investigator — Washington University School of Medicine in St Louis
Locations (5):
- United States (5):
  - Keck School of Medicine of the University of Southern California, Los Angeles, California
  - Fairview Health Services, Minneapolis, Minnesota
  - Washington University School of Medicine/St Louis Children's Hospital, St Louis, Missouri
  - Hearts for Hearing, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia - Buerger Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Data will be shared through presentations at relevant scientific meetings and through publication(s) in peer-reviewed journals. As required by the NIH Public Access Policy, an electronic version of final manuscripts resulting from this study will be submitted to the NIH National Library of Medicine PubMed Central (PMC) upon acceptance for publication. The few numbers of children at each study site who meet the inclusion criteria and receive a cochlear implant puts participant's privacy at risk if individual data are shared.